CLINICAL TRIAL: NCT00574080
Title: UARK 2006-15: A Phase III Randomized Study of Tandem Transplants With or Without Bortezomib (Velcade) and Thalidomide (Thalomid) to Evaluate Its Effect on Response Rate and Durability of Response in Multiple Myeloma Patients
Brief Title: UARK 2006-15: A Study of Tandem Transplants With or Without Bortezomib and Thalidomide
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-15
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — dexamethasone acetate; Neoadjuvant Therapy; Cytarabine; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): DPACE Induction, Melphalan/DPACE Transplant 1, BEAM Transplant 2, DPACE Consolidation, Dexamethasone Maintenance with Interim dexamethasone between treatment phases
  Interventions: Drug: Interim/Maintenance Dexamethasone; Drug: Induction/Consolidation Dexamethasone; Drug: Induction/Consolidation Cisplatin; Drug: Induction/Consolidation Adriamycin; Drug: InductionConsolidation Cyclophosphamide; Drug: Induction/Consolidation Etoposide; Drug: Induction Pegfilgrastim; Drug: Transplant 1 Dexamethasone; Drug: Transplant 1 Cisplatin; Drug: Transplant 1 Adriamycin; Drug: Transplant 1 Cyclophosphamide; Drug: Transplant 1 Etoposide; Drug: Transplant 1 Melphalan; Drug: Transplant 1 and 2 Pegfilgrastim; Procedure: Autologous Peripheral Blood Stem Cell Transplant (ASCT); Drug: Transplant 2 Carmustine; Drug: Transplant 2 Etoposide; Drug: Transplant 2 Cytarabine; Drug: Transplant 2 Melphalan; Drug: Transplant 2 Dexamethasone
- Arm B (Experimental): DPACE Induction, Melphalan/DPACE + VTD Transplant 1, BEAM + VTD Transplant 2, DPACE Consolidation, Dexamethasone Maintenance with Interim dexamethasone between treatment phases
  Interventions: Drug: Interim/Maintenance Dexamethasone; Drug: Induction/Consolidation Dexamethasone; Drug: Induction/Consolidation Cisplatin; Drug: Induction/Consolidation Adriamycin; Drug: InductionConsolidation Cyclophosphamide; Drug: Induction/Consolidation Etoposide; Drug: Induction Pegfilgrastim; Drug: Transplant 1 Dexamethasone; Drug: Transplant 1 Cisplatin; Drug: Transplant 1 Adriamycin; Drug: Transplant 1 Cyclophosphamide; Drug: Transplant 1 Etoposide; Drug: Transplant 1 Melphalan; Drug: Transplant 1 and 2 Pegfilgrastim; Procedure: Autologous Peripheral Blood Stem Cell Transplant (ASCT); Drug: Transplant 2 Carmustine; Drug: Transplant 2 Etoposide; Drug: Transplant 2 Cytarabine; Drug: Transplant 2 Melphalan; Drug: Transplant 2 Dexamethasone; Drug: Transplant 1 and 2 Bortezomib; Drug: Transplant 1 and 2 Thalidomide

INTERVENTIONS:
Drug: Interim/Maintenance Dexamethasone — 20 mg Days 1-4 every 3 weeks in the interim between treatment phases and during maintenance
  Other Names: Dex; Dexamethasone acetate
Drug: Induction/Consolidation Dexamethasone — 40 mg Days 1-4
  Other Names: Dex; Dexamethasone acetate
Drug: Induction/Consolidation Cisplatin — 10 mg/m2 by continuous infusion Days 1-4
Drug: Induction/Consolidation Adriamycin — 10 mg/m2 by continuous infusion Days 1-4
Drug: InductionConsolidation Cyclophosphamide — 400 mg/m2 by continuous infusion Days 1-4
Drug: Induction/Consolidation Etoposide — 40 mg/m2 by continuous infusion Days 1-4
Drug: Induction Pegfilgrastim — 6 mg Days 6 and 13
Drug: Transplant 1 Dexamethasone — 20 mg Days -4, -3, -2, -1 and +4, +5, +6, and +7
Drug: Transplant 1 Cisplatin — 20 mg/m2 by continuous infusion Days -3 and -2
Drug: Transplant 1 Adriamycin — 20 mg/m2 by continuous infusion Days -3 and -2
Drug: Transplant 1 Cyclophosphamide — 800 mg/m2 by continuous infusion Days -3 and -2
Drug: Transplant 1 Etoposide — 80 mg/m2 by continuous infusion Days -3 and -2
Drug: Transplant 1 Melphalan — 50 mg/m2 Days -2 and -1
Drug: Transplant 1 and 2 Pegfilgrastim — 6 mg Day +6
Procedure: Autologous Peripheral Blood Stem Cell Transplant (ASCT) — Day 0
Drug: Transplant 2 Carmustine — 300 mg/m2 Day -5
Drug: Transplant 2 Etoposide — 200 mg/m2 Days -5, -4, -3, -2
Drug: Transplant 2 Cytarabine — 400 mg/m2 Days -5, -4, -3, -2
  Other Names: Ara-C
Drug: Transplant 2 Melphalan — 140 mg/m2 Day -1
Drug: Transplant 2 Dexamethasone — 20 mg Days -5, -4, -3, -2, +4, +5, +6, +7
Drug: Transplant 1 and 2 Bortezomib — 1 mg/m2 Days -4, -1, +3, +7
  Other Names: Velcade
  Arms: Arm B
Drug: Transplant 1 and 2 Thalidomide — 200 mg Days -4 to +5
  Arms: Arm B

SUMMARY:
Add three drugs, bortezomib, thalidomide, and dexamethasone (VTD) to the high dose chemotherapy regimen immediately before transplant (DPACE/Melphalan) to try to improve myeloma response and acquire longer survival for participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic multiple myeloma, sensitive or refractory to at least one prior line of chemotherapy.
* Karnofsky performance score > 60%, unless due to MM.
* Patients must be <75 years of age at the time of registration.
* Patient must not have had a prior auto- or allotransplant.
* Patient must have signed an IRB-approved informed consent and understand the investigational nature of the study.
* Negative serology for HIV.
* Baseline biopsies and laboratory studies are to be completed within 35 days of registration, within 60 days for scans and radiological studies; patients must not have a history of severe chronic obstructive or chronic restrictive pulmonary disease. Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted. Patients unable to complete pulmonary function tests because of myeloma-related chest pain, must have a high resolution CT scan of the chest and must also have acceptable arterial blood gases defined as P02 greater than 70.
* Patients with recent (< 6 months) myocardial infarction, unstable angina, difficult to control congestive heart failure, uncontrolled hypertension, or difficult to control cardiac arrhythmias are ineligible. Ejection fraction by ECHO or MUGA must be > 40% and must be performed within 60 days prior to registration, unless the patient has received chemotherapy within that period of time (dexamethasone and thalidomide excluded), in which case the LVEF must be repeated.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years. Prior malignancy is acceptable provided there has been no evidence of disease within the three-year interval or if the malignancy is considered much less life threatening than the myeloma.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Patients must be able to receive full doses of D PACE, in the opinion of the treating investigator, with the exception that patients with creatinine clearance 30-50 ml/min will receive only 50% of the cisplatin dose.

Exclusion Criteria:

* Fever or active infection requiring intravenous antibiotic, defined as fever or antibiotics within 72 hours from baseline.
* Severe renal dysfunction, defined as a creatinine > 3mg/dl or a creatinine clearance of < 30ml/min.
* Significant neurotoxicity, defined as grade > 3 neurotoxicity per NCI Common Toxicity Criteria (See Appendix).
* Platelet count < 100,000/mm^3, or ANC < 1,000/μl
* POEMS Syndrome.
* Clinically significant hepatic dysfunction as noted by direct bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis.
* New York Hospital Association (NYHA) Class III or Class IV heart failure.
* Myocardial infarction within the last 6 months.
* Patients with a history of treatment for clinically significant ventricular cardiac arrhythmias.
* Poorly-controlled hypertension, diabetes mellitus, or other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Prior adriamycin exposure >450 mg/m^2
* Prior exposure to thalidomide which resulted in severe toxicity requiring drug discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are myeloma patients who have already received one or more treatment regimens and are seen at our facility
Groups:
- VTD + DPACE/Melphalan: Velcade, thalidomide, and dexamethasone + Dexamethasone, CisPlatin, Adriamycin, Cyclophosphamide, and Etoposide & Melphalan
- DPACE/Melphalan: Dexamethasone, CisPlatin, Adriamycin, Cyclophosphamide, and Etoposide & Melphalan
Period: Overall Study
Arm/Group | VTD + DPACE/Melphalan | DPACE/Melphalan
Started | 10 | 10
Completed | 0 | 0
Not Completed | 10 | 10
Not completed — Death | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VTD + DPACE/Melphalan | DPACE/Melphalan | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (5.01) | 59 (8.67) | 57.6 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival
Description: Time from study registration until disease progression or death.
Time Frame: Up to 3 years 8 months
Population: no analysis, participants either died or were withdrawn by PI. study terminated with <10% of target accrual enrolled.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | VTD + DPACE/Melphalan | DPACE/Melphalan
Serious Adverse Events (participants affected / at risk) | 4/10 | 3/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VTD + DPACE/Melphalan (N=10) | DPACE/Melphalan (N=10)
embolus (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
death (General disorders) | 1 (1) | 0 (0) — progressive disease
death (Cardiac disorders) | 0 (0) | 1 (1) — cardiac failure
death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — secondary malignancy
death (General disorders) | 2 (2) | 0 (0) — no cause listed
death (General disorders) | 0 (0) | 1 (1) — infection
death (General disorders) | 1 (1) | 0 (0) — sepsis

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects to be analyzed. Less than 10% of the target accrual were enrolled before termination of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes